CLINICAL TRIAL: NCT04005274
Title: Is Rate of Force Development (RFD) Superior to Isometric Strength (QS) of the Quadriceps as a Predictor of Functional Performance After Anterior Cruciate Ligament Reconstruction
Brief Title: Rate of Force Development vs Isometric Strength of Quadriceps
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: KPSC IRB 12068
Record Dates: First submitted 2019-06-20; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Post ACL Reconstruction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Peak isometric strength of quadriceps (QI) has been used to help determine an athletes ability to safely return back to sport following an anterior cruciate ligament (ACL) reconstruction surgery. However, rate of force development (RFD) of the quadriceps, or how fast the quadriceps are able to reach their peak strength, is rarely used as part of this decision despite the role it plays in protecting the knee. This retrospective data only study will look back at the limb symmetry index (LSI) of patients post ACL reconstruction for the Noyes Hop Test, QI, and RFD. The hypothesis is that RFD does not recover at the same rate as Noyes Hop Test and QI.

ELIGIBILITY:
Inclusion Criteria:

* No pain (at baseline) or edema/effusion
* Full knee range of motion
* Post Op: 20 weeks - 2 years
* Non antalgic gait

Exclusion Criteria:

* History of low back pain or other lower extremity injury within 1 year, skeletal immature, pregnant, concomitant ligament injury

Min Age: 14 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Kaiser Permanente patients attending out-patient physical therapy post ACL reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Limb Symmetry (Noyes hop testing, Isokinetic testing-rate of force development, Isokinetic testing-quadriceps index) | March - June 2019
  Limb symmetry was calculated comparing surgical leg over non-surgical leg giving a percentage. A percentage will be calculated for each one of the 3 observations allowing easy comparison with same unit of measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente West Los Angeles Medical Center, West Los Angeles, California, United States